CLINICAL TRIAL: NCT02542865
Title: Clinical Study to Measure the Impact of Fortified Malt Based Food on Immunity Outcomes in School Children
Brief Title: A Study to Investigate the Impact of Fortified Malt Based on Immunity Outcomes in School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 204477
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Results first posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-11

CONDITIONS: Growth and Development

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Group (Experimental): Fortified malt based food (27 grams) made up in 150 mL lukewarm water administered twice daily
  Interventions: Dietary Supplement: Fortified malt based food
- Control Group (No Intervention): No treatment was administered

INTERVENTIONS:
Dietary Supplement: Fortified malt based food — Fortified malt based food
  Arms: Test Group

SUMMARY:
This study will test the hypothesis that a fortified malt based food may improve immunity outcomes in 7-10 year old school age children.

DETAILED DESCRIPTION:
This will be a single centre, multiple sites, open label, two-arm, parallel-group, stratified by gender, matched pair cluster randomised, controlled study in children aged 7-10 years.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrates understanding of the study and willingness to participate as evidenced by the parent's and/or LAR's voluntary written informed consent as well as written assent by the child and has received a signed and dated copyof the informed consent form as well as the assent form.
* Boys and girls aged between 7-10 years
* Child and parent/LAR understand and are willing, able and likely to comply with all study procedures and restrictions.
* Good general and mental health with, in the opinion of the investigator or medically qualified designee: No clinically significant and relevant abnormalities in medical history or upon physical examination and absence of any condition that could affect the child's safety or wellbeing or their ability to understand and follow study procedures and requirements.
* Participants with HAZ of ≥-3 to ≤-1.

Exclusion Criteria:

* Children in Care (CiC): A child who has been placed under the control or protection of an agency, organisation, institution or entity by the courts, the government or a government body, acting in accordance with powers conferred on them by law or regulation. The definition of a CiC can include a child cared for by foster parents or living in a care home or institution, provided that the arrangement falls within the definition above. The definition of a CiC does not include a child who is adopted or has an appointed legal guardian.
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Indication that child is likely to move out of geographical range of the study within the period of study intervention and activities, thus hindering the child's compliance to study activities.
* Clinical Study/Experimental Medication: a) Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit, participation in any nutritional study or didactic nutrition education in the last 6 months of the screening visit and previous participation in this study.
* Child with severe anaemia (Hemoglobin <8g/dL).
* Children with history of use of immunosuppressive therapy e.g. oral corticosteroids or chemotherapy in past six months prior to the screening visit.
* Current or relevant history of any serious, severe or unstable physical or psychiatric illness or any medical disorder that would make the participant unlikely to fully complete the study or any condition that presents undue risk from the test product or procedures, on the discretion of study physician.
* Recent history [2 months] of serious infections, injuries and/ or surgeries in the opinion of the investigator.
* Children consuming nutritional supplements and/or health food drinks on a regular basis (≥3 times a week) in last 3 months.
* Child belonging to an employee of the sponsor or the study site or members of their immediate family or sibling of a child already enrolled in the study.

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 924 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2018-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Pune, India

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 4 schools in India.
Pre-assignment Details: Total 958 participants were screened. Of these, 924 participants were enrolled for randomized treatment, of which, 2 participants withdrew their consent before starting the treatment. 34 participants were not enrolled, of which, 11 did not meet study criteria, 22 had withdrawal of consent and 1 identified as screen failure.
Groups:
- Fortified Malt Based Food Plus Dietary Counselling: In this group, participants received fortified malt based food, 27 grams (g) powder made up in 150 milliliters (mL) lukewarm water, twice daily (during school days first dose was given as soon as the participants entered the school and the second dose just prior to school dismissal and during holidays, first dose was provided in the morning and the second dose administered in the evening, by parents/LARs [legally acceptable representative]) for 9 months. Dietary counseling was provided to both participants and parents/LARs separately in 2 mandatory sessions, which were followed up in 5 follow up sessions.
- Dietary Counselling Only: In this group, only dietary counseling was provided to both participants and parents/LAR. This was matched to test group (fortified malt based product plus dietary counselling) with respect to quality, content and duration.
Period: Overall Study
Arm/Group | Fortified Malt Based Food Plus Dietary Counselling | Dietary Counselling Only
Started (Participants randomized to the treatment arms) | 462 | 462
Treated (2 participants withdrew their consent before starting the treatment.) | 460 | 462
Completed | 445 | 462
Not Completed | 17 | 0
Not completed — Identified as screen failure | 1 | 0
Not completed — Withdrawal by Subject | 16 | 0

BASELINE CHARACTERISTICS:
Population: Baseline assessment was performed on Safety Population (N=922) which included all randomized participants who received at least 1 dose of study treatment. The safety population was based on the product the participant was planned to receive.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fortified Malt Based Food Plus Dietary Counselling | Dietary Counselling Only | Total
Number analyzed (Participants) | 460 | 462 | 922
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.0 (0.78) | 7.9 (0.84) | 8.0 (0.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 196 | 206 | 402
  Male | 264 | 256 | 520
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 460 | 462 | 922
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: Centimeters (cm)] | 120.83 (4.804) | 120.71 (5.070) | 120.77 (4.937)
Weight [Median (Standard Deviation); unit: Kilograms (kg)] | 22.66 (4.053) | 22.14 (4.565) | 22.40 (4.323)

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Ill Days Due to Gastrointestinal (GI) and Respiratory Illness at Month 9
Description: Number of days a participant was ill due to GI and/or respiratory illness as diagnosed by physician, as per criteria defined, over the intervention duration. This equals total number of days (symptomatic or asymptomatic) in illnesses episodes whereas each episode is defined as an incidence of illness followed by at least 3 symptoms free days. GI illness was defined as an acute illness that includes any of following symptoms:3 or more loose/liquid/watery stools and/or vomiting in 24hours (h). Respiratory illness was defined as an acute illness that included more than or equal to [>=] 1 of the following symptoms: runny nose, stuffy or blocked nose, cough fever or chills, sore throat or sneezing.
Time Frame: At month 9
Population: mITT (modified intent-to-treat) population (N=907) included all treated participants with post-treatment assessments who completed the entire study of 9 months.
Measure: Mean (Standard Deviation); unit: Number of days
Arm/Group | Fortified Malt Based Food Plus Dietary Counselling | Dietary Counselling Only
Number analyzed (Participants) | 445 | 462
Number of days | 2.3 (5.23) | 8.2 (7.97)
Statistical Analysis 1: Comparison: Fortified Malt Based Food Plus Dietary Counselling vs Dietary Counselling Only; Test type: Superiority; p = 0.0628, ANCOVA; Analysis of variance(ANCOVA):cluster/school=random effect,product group and gender=fixed effects,baseline Individual Dietary Diversity Score=covariate; Mean Difference (Net) = -6.0, 95% CI 2-sided [-12.7 to 0.8], Standard Error of Mean 1.56 — Difference is difference in back-transformed adjusted means for Test Group (fortified malt based food plus dietary counselling) minus Control Group (dietary counselling only)
Statistical Analysis 2: Comparison: Fortified Malt Based Food Plus Dietary Counselling vs Dietary Counselling Only; Since the distribution of the data was found to be more skewed with more zero counts than was anticipated at the time the trial was designed, an additional analysis of log (+1)-transformed data was performed; Test type: Superiority; p = 0.0390, ANCOVA; ANCOVA:cluster/school=random effect,product group and gender=fixed effects,baseline Individual Dietary Diversity Score=covariate; Mean Difference (Net) = -4.9 — Difference is difference in back-transformed adjusted means for Test Group minus Control Group. The corresponding CI is not presented as there is no direct back-transformation

2. Secondary Outcome: Frequency of GI and Respiratory Illnesses at Month 9
Description: Number of episodes of GI and respiratory illnesses was calculated at month 9 using a diagnosis form (DF) which were used to note the diagnosis, severity, and school absenteeism due to GI and respiratory illnesses only, as defined in the study protocol. The DF captured the start and end date of all occurrences of GI and respiratory illnesses in the week. The frequency was calculated as total number of GI and respiratory illness episodes, divided by duration of intervention, where each episode is defined as each incidence of illness followed by at least uninterrupted 3 symptom free days. Therefore, the formula for calculation used was: frequency (per month) = number of episodes multiply (x) 30 and divided by (/) number of days between first and last visit.
Time Frame: At month 9
Population: mITT population (N=907) included all treated participants with post-treatment assessments who completed the entire study of 9 months.
Measure: Mean (Standard Deviation); unit: Number of episodes per month
Arm/Group | Fortified Malt Based Food Plus Dietary Counselling | Dietary Counselling Only
Number analyzed (Participants) | 445 | 462
Number of episodes per month | 0.067 (0.1100) | 0.241 (0.1584)

3. Secondary Outcome: Severity of GI Illnesses at Month 9
Description: Severity of GI illness was calculated at month 9 using DF with observations listed by study physician based on assessment of severity grade: classified as, diarrhea (Mild, increase of less than [<] 4 stools per [/] day over baseline; Moderate, increase of 4 to 6 stools/day over baseline; Severe, increase of more than or equal to [>=]7 loose stools/day over baseline) and vomiting (1-2 episodes, separated by 5 minutes[min] in 24 h; Moderate, 3-5 episodes, separated by 5 min in 24 h; Severe, >=6 episodes, separated by 5 min in 24 h. The count of participants was calculated based on the episode of worst severity. Lower severity indicates no illness of participant.
Time Frame: At month 9
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fortified Malt Based Food Plus Dietary Counselling | Dietary Counselling Only
Number analyzed (Participants) | 445 | 462
Participants
  Mild | 30 | 163
  Moderate | 13 | 20
  Severe | 0 | 0
  No illness | 402 | 279

4. Secondary Outcome: Severity of Respiratory Illnesses at Month 9
Description: Intensity of respiratory illness was calculated at month 9 using DF with observations listed by study physician based on assessment of severity grade classified as, Mild or Grade1 is asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated; Moderate or Grade 2 is minimal, local or non-invasive intervention indicated; limiting age-appropriate instrumental activities of daily living (ADL). Instrumental ADL refer to school attendance, playing, studying, participating in school activities; and Severe or Grade 3 and 4: Grade 3 is severe or medically significant, but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL. Self-care ADL refers to bathing, dressing and undressing, feeding self, using the toilet, taking medications, and not bedridden; Grade 4 is life-threatening consequences; urgent indication indicated.
Time Frame: At month 9
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Fortified Malt Based Food Plus Dietary Counselling | Dietary Counselling Only
Number analyzed (Participants) | 445 | 462
Participants
  Mild | 97 | 293
  Moderate | 50 | 89
  Severe | 12 | 8
  No illness | 286 | 72

5. Secondary Outcome: School Absenteeism Assessment Due to GI and Respiratory Illnesses at Month 9
Description: School absenteeism was calculated as number of days when a participant failed to attend school because of GI and/or respiratory illnesses. DF was used to note school absenteeism , however it was marked for absenteeism due to GI and respiratory illnesses only.
Time Frame: At month 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Number of days
Arm/Group | Fortified Malt Based Food Plus Dietary Counselling | Dietary Counselling Only
Number analyzed (Participants) | 445 | 462
Number of days | 0.1 (0.61) | 0.6 (1.34)

6. Secondary Outcome: Change From Baseline in Body Mass Index (BMI) at Month 9
Description: Change in Body Mass Index (BMI) was calculated at month 9 using anthropometric measurements. For measuring participant's height, portable stadio-meter was used with the participant standing barefoot; to the nearest 0.1 centimeters (cm) and average of 3 measurements were recorded. All data recorded in cm were converted to meters (m) for BMI calculation. For measuring participant's weight, standardized weighing scale was used in standard clothing to the nearest 0.1kilograms (kg) and average of 3 measurements were recorded. BMI value was calculated using the formula weight divided by square of height (weight [kilogram (kg)/ Height [meter (m)]^2)
Time Frame: At screening and month 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kilograms per meter square (kg/m^2)
Arm/Group | Fortified Malt Based Food Plus Dietary Counselling | Dietary Counselling Only
Number analyzed (Participants) | 445 | 462
Kilograms per meter square (kg/m^2)
  At month 9 | 15.668 (2.3446) | 15.187 (2.3620)
  Change from baseline at month 9 | 0.194 (0.9948) | 0.068 (1.4408)

7. Secondary Outcome: Change From Baseline in Gut Integrity/ Health Measured by Urine Lactulose: Mannitol Test at Month 9
Description: Improvement in gut wall integrity was considered a possible factor to assess the micronutrient absorption. Lactulose mannitol test was used to evaluate change in gut wall permeability status to assess impact on micronutrient absorption. After 3h of fasting, pre-measured amount of lactulose/mannitol solution (2 milliliter/Kilogram [mL/Kg] of body weight) containing lactulose (250 milligram/milliliter [mg/mL])] and mannitol (50 mg/mL) was administered as a test solution. Participants were allowed to return to their regular diet 30 minutes after ingestion of the test solution. During the 2.5 h time, participants were offered liquids frequently in order to permit collection of an adequate volume of urine. After 2.5 h, urine collection was performed. All urine passed over duration of 2.5 h was collected and analysed. High Performance Liquid Chromatography (HPLC) test method was used to measure the levels. The normal range of urinary lactulose: mannitol is less than [<] 0.035.
Time Frame: At baseline and month 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio (unitless)
Arm/Group | Fortified Malt Based Food Plus Dietary Counselling | Dietary Counselling Only
Number analyzed (Participants) | 445 | 462
Ratio (unitless)
  At baseline: number analyzed (Participants) | 431 | 452
  At baseline | 0.0504 (0.19891) | 0.0218 (0.01150)
  At month 9: number analyzed (Participants) | 430 | 440
  At month 9 | 0.0429 (0.06399) | 0.0405 (0.12221)
  Change from baseline at month 9: number analyzed (Participants) | 416 | 431
  Change from baseline at month 9 | -0.0082 (0.21151) | 0.0192 (0.12400)

8. Secondary Outcome: Change From Baseline in Gut Integrity/ Health Using Urinary Neopterin Assessment at Month 9
Description: Improvement in gut wall integrity was considered a possible factor to assess the micronutrient absorption. Neopterin test was used to evaluate change in gut wall permeability status to assess impact on micronutrient absorption. Spontaneous random urine was collected from the participants and a volume of 2mL per participant was stored and analysed. Urine sample for this test were collected prior to administration of Lactulose/Mannitol solution. Enzyme-linked immunosorbent assay (ELISA) test method was used to measure the levels. The values were measured in Millimoles per moles of creatinin (mmol/mol creatinin). The normal range of urinary neopterin is 0.10-5.00 mmol/ mol creatinin.
Time Frame: At baseline and month 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/mol creatinin
Arm/Group | Fortified Malt Based Food Plus Dietary Counselling | Dietary Counselling Only
Number analyzed (Participants) | 445 | 462
mmol/mol creatinin
  At baseline | 0.419 (0.3967) | 0.388 (0.4410)
  At month 9 | 0.537 (0.4955) | 0.557 (0.4937)
  Change from baseline at month 9 | 0.119 (0.6188) | 0.169 (0.6302)

9. Secondary Outcome: Change From Baseline in Mucosal Immunity Using Salivary Immunoglobulin A (IgA) Assessment at Month 9
Description: Quantity of salivary IgA was used to measure the impact of fortified malt based food on mucosal immunity. Saliva was collected using saliva collection aid (SCA). Ribbed-end of the SCA were securely placed into a pre-labeled collection vial. Participants were instructed to pool the saliva in mouth. SCA was placed on mouth entry. Then, participants were asked to tilt the head forward, and gently force saliva through the SCA into the vial to fill with at least 50 microliters (mcL) of volume. A small amount of air space was reserved in the vial to accommodate liquid expansion during freezing. After collection of sample, SCA was removed and discarded and cap was attached to collection vial and tightened. ELISA test method was used to detect the salivary IgA levels. The normal range of salivary IgA is 25.00-168.00 milligrams per liter (mg/L).
Time Frame: At baseline and month 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Fortified Malt Based Food Plus Dietary Counselling | Dietary Counselling Only
Number analyzed (Participants) | 445 | 462
mg/L
  At baseline | 84.659 (33.7306) | 79.278 (33.3108)
  At month 9 | 94.392 (29.3311) | 90.386 (29.2448)
  Change from baseline at month 9 | 9.733 (25.7247) | 11.108 (24.9461)

10. Secondary Outcome: Change From Baseline in Serum Levels of Micronutrient Vitamin A and Trace Elements Zinc (Zn), Copper (Cu) and Iron (Fe) at Month 9
Description: Quantity of micronutrients, serum vitamin-A and of trace elements Zn, Cu and Fe levels in serum were used to assess the impact of fortified malt based food product on nutrient biochemistry at month 9. To quantitate the nutrient biochemistry, a total volume of approximately 14 milliliters (ml), 7ml each at screening and at month 9, whole blood sample was collected from each participant after application of an anesthetic patch/ointment. The test methods used were ELISA for vitamin-A and colorimetric assays for Zn, Cu and Fe as 5-Br-PAPS; 3,5-Dibromo-PAES and TPTZ, respectively. The normal range of serum Vitamin-A is 26.00-49.00 micrograms per deciliter (mcg/dL) and serum Zn is 78.00-105.00 (male and females aged 7-9 years), 78.00- 118.00 (females aged 10 years) and 78.00-98.00 (males aged 10 years) mcg/dL. The normal range of serum Cu is 51.00-121.00 mcg/dL and serum Fe is 50.00-120.00 mcg/dL.
Time Frame: At baseline and month 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/dL
Arm/Group | Fortified Malt Based Food Plus Dietary Counselling | Dietary Counselling Only
Number analyzed (Participants) | 445 | 462
mcg/dL
  Serum Vitamin-A : at baseline | 29.522 (6.3004) | 28.141 (5.4046)
  Serum Vitamin-A : at month 9 | 31.631 (7.4251) | 31.446 (6.5425)
  Serum Vitamin-A : change from baseline at month 9 | 2.109 (8.0874) | 3.305 (7.4460)
  Serum Zn: at baseline | 72.166 (19.8017) | 72.583 (19.9806)
  Serum Zn: at month 9 | 88.795 (22.4039) | 89.450 (23.1540)
  Serum Zn: change from baseline at month 9 | 16.629 (19.8966) | 16.867 (19.6339)
  Serum Cu: at baseline | 117.896 (15.9230) | 117.771 (16.0825)
  Serum Cu: at month 9 | 116.514 (19.2957) | 116.996 (18.0636)
  Serum Cu: change from baseline at month 9 | -1.382 (19.0421) | -0.775 (19.3061)
  Serum Fe: at baseline | 70.087 (29.7686) | 71.426 (29.1396)
  Serum Fe: at month 9 | 70.843 (23.5478) | 70.349 (21.7732)
  Serum Fe: change from baseline at month 9 | 0.755 (27.2156) | -1.077 (24.7602)

11. Secondary Outcome: Change From Baseline in Serum Levels of Trace Element Selenium (Se) at Month 9
Description: Quantity of the trace element, serum Se was used to assess the impact of fortified malt based food product on nutrient biochemistry at month 9. To quantitate the nutrient biochemistry, a total volume of approximately 14 milliliters (ml), 7ml each at screening and at month 9, whole blood sample was collected from each participant after application of an anesthetic patch/ointment. The test method used was inductively coupled plasma mass spectrometry (ICP-MS). The normal range of serum Se is 55.00-134.00 micrograms per liter (mcg/L).
Time Frame: At baseline and month 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mcg/L
Arm/Group | Fortified Malt Based Food Plus Dietary Counselling | Dietary Counselling Only
Number analyzed (Participants) | 445 | 462
mcg/L
  Serum Selenium: at baseline | 83.625 (12.6082) | 85.905 (12.2420)
  Serum Selenium: at month 9 | 92.703 (17.5743) | 91.286 (17.0242)
  Serum Selenium: change from baseline at month 9 | 9.078 (17.2151) | 5.381 (17.0555)

12. Secondary Outcome: Change From Baseline in Serum Levels of Micronutrient Vitamin B12 at Month 9
Description: Quantity of micronutrient, serum vitamin-B12 was used to assess the impact of fortified malt based food product on nutrient biochemistry at month 9. To quantitate the nutrient biochemistry, a total volume of approximately 14 milliliters (ml), 7ml each at screening and at month 9, whole blood sample was collected from each participant after application of an anesthetic patch/ointment. The test method ELISA was used to measure the levels. The normal range of the serum vitamin B12 is 312.00-1237.00 is picograms per milliliter (pg/mL).
Time Frame: At baseline and month 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Fortified Malt Based Food Plus Dietary Counselling | Dietary Counselling Only
Number analyzed (Participants) | 445 | 462
pg/mL
  At baseline | 374.384 (87.3163) | 375.671 (97.5075)
  At month 9 | 429.682 (85.4784) | 419.310 (91.2245)
  Change from baseline at month 9 | 55.299 (80.1776) | 43.638 (78.1703)

13. Secondary Outcome: Change From Baseline in Serum Levels of Micronutrients Vitamin-D and Serum Folate at Month 9
Description: Quantity of serum vitamin-D (25-hydroxycholecalciferol) and serum folate micronutrients were used to assess the impact of fortified malt based food product on nutrient biochemistry at month 9. To quantitate the nutrient biochemistry, a total volume of approximately 14 milliliters (ml), 7ml each at screening and at month 9, whole blood sample was collected from each participant after application of an anesthetic patch/ointment. The test method ELISA was used to measure the levels. The normal range of serum Vitamin-D is 30.00-100.00 nanograms per milliliter (ng/mL) and serum folate is 5.00-21.00 ng/mL.
Time Frame: At baseline and month 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Fortified Malt Based Food Plus Dietary Counselling | Dietary Counselling Only
Number analyzed (Participants) | 445 | 462
ng/mL
  Serum Vitamin-D: at baseline | 17.479 (5.6318) | 17.893 (5.1043)
  Serum Vitamin-D: at month 9 | 20.329 (5.7833) | 20.054 (5.0556)
  Serum Vitamin-D: change in baseline at month 9 | 2.850 (4.9529) | 2.161 (4.8962)
  Serum folate: at baseline | 4.510 (0.7322) | 4.415 (0.7075)
  Serum folate: at month 9 | 5.171 (0.7914) | 5.070 (0.8106)
  Serum folate: change from baseline at month 9 | 0.661 (0.7897) | 0.656 (0.7631)

14. Secondary Outcome: Change From Baseline in Serum Levels of Micronutrient Vitamin-E at Month 9
Description: Quantity of micronutrient, serum vitamin-E was used to assess the impact of fortified malt based food product on nutrient biochemistry at month 9. To quantitate the nutrient biochemistry, a total volume of approximately 14 milliliters (ml), 7ml each at screening and at month 9, whole blood sample was collected from each participant after application of an anesthetic patch/ointment. The test method ELISA was used to measure the levels. The normal range of serum vitamin-E is 0.30-0.90 milligrams per deciliter (mg/dL).
Time Frame: At baseline and month 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Fortified Malt Based Food Plus Dietary Counselling | Dietary Counselling Only
Number analyzed (Participants) | 445 | 462
mg/dL
  At baseline | 0.493 (0.1435) | 0.475 (0.1616)
  At month 9 | 0.541 (0.1407) | 0.494 (0.1145)
  Change from baseline at month 9 | 0.048 (0.1549) | 0.018 (0.1452)

15. Secondary Outcome: Change From Baseline in Serum Levels of Ferritin Using Blood Testing at Month 9
Description: Quantitative analysis of serum ferritin was studied to measure iron status. Its value was adjusted by other acute phase proteins such as C-reactive protein (CRP) and Alpha 1-acid glycoprotein (AGP) which are not related to iron status and played a role as a part of assessment on inflammatory status and to adjust ferritin status. To quantitate this load, a total volume of approximately 14 milliliters (ml), 7ml each at screening and at month 9, whole blood sample was collected from each participant after application of an anesthetic patch/ointment. The turbidimetry test method was used to measure the levels.The normal range of serum ferritin is 7.00-140.00 nanograms per milliliter (ng/ml).
Time Frame: At baseline and month 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Fortified Malt Based Food Plus Dietary Counselling | Dietary Counselling Only
Number analyzed (Participants) | 445 | 462
ng/ml
  At baseline | 24.261 (18.3705) | 22.743 (13.5996)
  At month 9 | 27.239 (12.7525) | 25.223 (13.6193)
  Change from baseline at month 9 | 2.978 (19.4921) | 2.480 (16.1006)

16. Secondary Outcome: Change From Baseline in Levels of Serum Transferrin Receptor (sTfR) Using Blood Testing at Month 9
Description: Quantitative analysis of sTfR along with serum iron and serum ferritin was studied to measure iron status. In cases of a high prevalence of infection and inflammation, sTfR becomes the choice of iron status marker. To quantitate this load, a total volume of approximately 14 milliliters (ml), 7ml each at screening and at month 9, whole blood sample was collected from each participant after application of an anesthetic patch/ointment. The immunoturbidimetry test method was used to measure the levels. The normal range of sTfR is 1.90-4.40 milligrams per liter (mg/L).
Time Frame: At baseline and month 9
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Fortified Malt Based Food Plus Dietary Counselling | Dietary Counselling Only
Number analyzed (Participants) | 445 | 462
mg/L
  At baseline | 1.564 (0.5009) | 1.521 (0.4937)
  At month 9 | 1.510 (0.3670) | 1.471 (0.3483)
  Change from baseline at month 9 | -0.055 (0.4181) | -0.050 (0.3594)

17. Secondary Outcome: Change From Baseline in Serum Levels of C-reactive Protein (CRP) and Alpha 1-acid Glycoprotein (AGP) Using Blood Testing at Month 9
Description: Quantitative analysis of acute phase proteins such as serum CRP and serum AGP were studied to assess inflammatory status and adjust ferritin status. To quantitate this load, a total volume of approximately 14 milliliters (ml), 7ml each at screening and at month 9, whole blood sample was collected from each participant after application of an anesthetic patch/ointment. The immunoturbidimetry test method was used to measure the levels of CRP and turbidimetry for AGP. The normal range of the serum CRP is less than (<) 0.50 milligrams per deciliter (mg/dL) and serum AGP is 50.00-120.00 mg/dL.
Time Frame: At baseline and month 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Fortified Malt Based Food Plus Dietary Counselling | Dietary Counselling Only
Number analyzed (Participants) | 445 | 462
mg/dL
  CRP: at baseline | 0.057 (0.1978) | 0.046 (0.1466)
  CRP: at month 9 | 0.114 (0.2117) | 0.103 (0.1839)
  CRP: change from baseline at month 9 | 0.058 (0.2682) | 0.057 (0.1916)
  AGP: at baseline | 74.888 (20.4840) | 74.542 (18.0323)
  AGP: at month 9 | 74.972 (18.8386) | 74.219 (16.9083)
  AGP: change from baseline at month 9 | 0.083 (18.8226) | -0.323 (16.7025)

18. Secondary Outcome: Change From Baseline in Individual Dietary Diversity Score (IDDS) at Month 9
Description: IDDS-measure of nutritional quality of individual's diet-assessed by questionnaire based on Guidelines for measuring household and individual dietary diversity set by Food and Agriculture Organisation (FAO) of United Nations[FAO guidelines dietary diversity,2011].Based on data of foods and beverages consumed in last 24h as captured by 24h dietary survey,appropriate food groups were selected. IDDS was calculated by adding number of food groups consumed by child over 24h recall period. Scoring 0-9with 1 point for foods that were consumed from each of food groups in previous 24h:starchy staples,dark green leafy vegetables,other vitamin A rich fruits and vegetables,other fruits and vegetables,organ meat, meat and fish, eggs, legumes, nuts, and seeds, milk and milk products. Based on IDDS,participants were listed into 3 food groups: a) less than or equal to [<=]3-low dietary diversity (DD);b)4-5-medium DD;c) greater than or equal to [>=]6-high DD. High score indicates nutrition rich food.
Time Frame: At baseline and month 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Diversity score
Arm/Group | Fortified Malt Based Food Plus Dietary Counselling | Dietary Counselling Only
Number analyzed (Participants) | 445 | 462
Diversity score
  At baseline | 4.2 (0.71) | 4.4 (0.67)
  At month 9 | 5.7 (1.23) | 4.6 (0.76)
  Change from baseline at month 9 | 1.5 (1.54) | 0.3 (0.99)

19. Secondary Outcome: Change From Baseline in Protein, Carbohydrates and Fat Consumption at Month 9
Description: Quantity of dietary intake was measured by protein, carbohydrate, and fat intake which was assessed from 24h dietary recall form. A structured interview was conducted based on a questionnaire. Parent/LARs provided the majority of information, with the child/ participant making additions to fill in the gaps. Both participants and parents/LARs recalled all food and beverage consumed by the child during previous 24h and information such as list and amount of ingredients, cooking method and portion size was recorded. Calculation on energy, protein, carbohydrates and fat were made using Dietsoft software based on Indian data (NIN [National Institute of Nutrition] and ICMR [Indian Council of Medical Research]) was used.
Time Frame: At baseline and month 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Grams (g)
Arm/Group | Fortified Malt Based Food Plus Dietary Counselling | Dietary Counselling Only
Number analyzed (Participants) | 445 | 462
Grams (g)
  Protein: at baseline | 38.840 (11.8775) | 42.406 (13.3945)
  Protein: at month 9 | 46.556 (11.7492) | 38.341 (11.0772)
  Protein: change from baseline at month 9 | 7.716 (17.3205) | -4.065 (16.5706)
  Carbohydrate: at baseline | 189.478 (50.7510) | 202.385 (55.0813)
  Carbohydrate: at month 9 | 186.223 (42.4576) | 181.126 (47.6042)
  Carbohydrate: change from baseline at month 9 | -3.255 (67.6676) | -21.259 (74.4880)
  Fat: at baseline | 47.516 (16.5686) | 40.034 (16.4056)
  Fat: at month 9 | 59.006 (18.0862) | 40.210 (16.2262)
  Fat: change from baseline at month 9 | 11.490 (23.3769) | 0.175 (20.6106)

20. Secondary Outcome: Change From Baseline in Energy Consumption at Month 9
Description: Quantity of dietary intake was also measured by energy intake which was assessed from 24-h dietary recall survey. A structured interview was conducted based on a questionnaire. Parent/LARs (legally appropriate representative) provided the majority of information, with the child making additions to fill in the gaps. Parents/LARs recalled all food and beverage consumed by the child during previous 24-h and information such as list and amount of ingredients, cooking method and portion size was recorded. Calculation on energy, protein, carbohydrates and fat were made using Dietsoft software based on Indian data (NIN and ICMR) was used.
Time Frame: At baseline and month 9
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Kilocalories (Kcal)
Arm/Group | Fortified Malt Based Food Plus Dietary Counselling | Dietary Counselling Only
Number analyzed (Participants) | 445 | 462
Kilocalories (Kcal)
  At baseline | 1395.142 (305.7777) | 1406.079 (352.7524)
  At month 9 | 1496.411 (299.0027) | 1309.889 (325.2896)
  Change from baseline at month 9 | 101.269 (446.1953) | -96.190 (484.0124)

ADVERSE EVENTS:
Time Frame: From baseline up to 9 months
Description: The Safety Population (N=922) included all participants who received at least 1 dose of the study product (test or reference product). Adverse Events (AEs) were regarded as treatment-emergent if they occurred on or after the first study product administration. If this date was missing, a suitable alternative was used for example a date of particular visit. All other AEs prior to this were considered non-treatment emergent.
Arm/Group | Fortified Malt Based Food Plus Dietary Counselling | Dietary Counselling Only
All-Cause Mortality (participants affected / at risk) | 0/460 | 0/462
Serious Adverse Events (participants affected / at risk) | 0/460 | 0/462
Other Adverse Events (participants affected / at risk) | 214/460 | 435/462
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fortified Malt Based Food Plus Dietary Counselling (N=460) | Dietary Counselling Only (N=462)
Diarrhea (Gastrointestinal disorders) | 21 (25) | 47 (52)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 6 (6) | 84 (99)
Malabsorption (Gastrointestinal disorders) | 18 (18) | 16 (16)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Post-tussive vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 13 (14) | 56 (59)
Pyrexia (General disorders) | 32 (35) | 49 (59)
Multiple allergies (Immune system disorders) | 0 (0) | 2 (2)
Seasonal allergy (Immune system disorders) | 0 (0) | 3 (3)
Bronchitis (Infections and infestations) | 1 (1) | 14 (14)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1)
Diarrhea infectious (Infections and infestations) | 1 (1) | 0 (0)
Gastritis viral (Infections and infestations) | 1 (1) | 2 (2)
Gastroenteritis (Infections and infestations) | 14 (16) | 32 (33)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 16 (18)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 8 (9)
Respiratory tract infection (Infections and infestations) | 10 (10) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 14 (15) | 115 (172)
Upper respiratory tract infection (Infections and infestations) | 116 (174) | 292 (542)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 4 (4) | 7 (7)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Skin abrasion (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood iron decreased (Investigations) | 0 (0) | 1 (1)
Blood zinc decreased (Investigations) | 0 (0) | 1 (1)
Transferrin decreased (Investigations) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2)
Allergic bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (4)
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 23 (27)
Allergic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 9 (11)
Allergic respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (16) | 28 (29)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 13 (14)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (5)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 75 (88)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 11 (11)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-10-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT02542865/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-02): https://cdn.clinicaltrials.gov/large-docs/65/NCT02542865/SAP_001.pdf